CLINICAL TRIAL: NCT00073853
Title: A Phase II Multicenter, Randomized-Controlled Study to Evaluate the Safety and Efficacy of Autologous Incubated Macrophages for the Treatment of Patients With Complete Spinal Cord Injuries
Brief Title: Autologous Incubated Macrophages for Patients With Complete Spinal Cord Injuries
Status: Suspended | Phase: Phase 2 | Type: Interventional
Sponsor: Proneuron Biotechnologies (Industry)
Collaborators: The Marcus Foundation (Other); B.I.R.D. (Israel-U.S. Binational Industrial Research and Development) (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-P-01
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2006-03

CONDITIONS: Spinal Cord Injury
Keywords: paraplegia; quadraplegia; tetraplegia; paralysis; nerve regeneration; Acute, Complete SCI
MeSH Terms: conditions — Spinal Cord Injuries; Paraplegia; Quadriplegia; Paralysis | interventions — Cell- and Tissue-Based Therapy

INTERVENTIONS:
Procedure: Autologous Incubated Macrophages (cell therapy)

SUMMARY:
Autologous Incubated Macrophages (ProCord) is being developed as a therapy for acute, complete spinal cord injury (SCI). The therapy is intended to reverse the loss of motor and sensory function.

Following non-CNS tissue injury, macrophages quickly arrive on the scene, where they clean up cell debris, secrete different molecules thus promoting a controlled inflammatory reaction that forms the first phase of the wound healing process. While this process occurs in most tissues, including peripheral nerves, it does not occur in the CNS, where macrophages and other immune cells are relatively rare, and their activities curtailed by a biochemical mechanism known as "immune privilege."

In animal studies, it appears that incubated macrophages circumvent the immune privilege, thus supporting the regrowth of axons through the injury site and enabling the recovery of neurological function. The concept derives from the pioneering research of Prof. Michal Schwartz at the Weizmann Institute of Science.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic SCI during last 14 days
* Age 16 to 65 years
* Complete spinal cord injury (ASIA A)
* Neurological level : C5 to T11
* MRI showing lesion

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Coma or other severe injury or disease
* Penetrating injury
* Ongoing mechanical ventilation
* Unsuitable based on MRI or other factor

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61
Dates: Start 2003-09

PRIMARY OUTCOMES:
Improvement of ASIA grade

SECONDARY OUTCOMES:
Sensory scores
Motor scores
Bladder and bowel function

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lammertse, M.D., Study Director — Craig Hospital; Nachshon Knoller, M.D., Study Director — Chaim Sheba Medical Center; Marca Sipski, M.D., Study Director — University of Miami; Edward Benzel, M.D., Study Director — The Cleveland Clinic
Locations (7):
- United States (6):
  - Craig Hospital, Englewood, Colorado
  - Shepherd Center, Atlanta, Georgia
  - UMDNJ, Newark, New Jersey
  - Kessler Medical Rehabilitation Research and Education Corporation, West Orange, New Jersey
  - Mount Sinai Spinal Cord Injury Model System, New York, New York
  - Shriners Hospital for Children, Philadelphia, Pennsylvania
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Knoller N, Auerbach G, Fulga V, Zelig G, Attias J, Bakimer R, Marder JB, Yoles E, Belkin M, Schwartz M, Hadani M. Clinical experience using incubated autologous macrophages as a treatment for complete spinal cord injury: phase I study results. J Neurosurg Spine. 2005 Sep;3(3):173-81. doi: 10.3171/spi.2005.3.3.0173. PMID 16235699
- [Background] Bomstein Y, Marder JB, Vitner K, Smirnov I, Lisaey G, Butovsky O, Fulga V, Yoles E. Features of skin-coincubated macrophages that promote recovery from spinal cord injury. J Neuroimmunol. 2003 Sep;142(1-2):10-6. doi: 10.1016/s0165-5728(03)00260-1. PMID 14512160
- [Background] Rapalino O, Lazarov-Spiegler O, Agranov E, Velan GJ, Yoles E, Fraidakis M, Solomon A, Gepstein R, Katz A, Belkin M, Hadani M, Schwartz M. Implantation of stimulated homologous macrophages results in partial recovery of paraplegic rats. Nat Med. 1998 Jul;4(7):814-21. doi: 10.1038/nm0798-814. PMID 9662373
- [Derived] Lammertse DP, Jones LA, Charlifue SB, Kirshblum SC, Apple DF, Ragnarsson KT, Falci SP, Heary RF, Choudhri TF, Jenkins AL, Betz RR, Poonian D, Cuthbert JP, Jha A, Snyder DA, Knoller N. Autologous incubated macrophage therapy in acute, complete spinal cord injury: results of the phase 2 randomized controlled multicenter trial. Spinal Cord. 2012 Sep;50(9):661-71. doi: 10.1038/sc.2012.39. Epub 2012 Apr 24. PMID 22525310